CLINICAL TRIAL: NCT05073991
Title: Incidence of Perioperative Mortality and Major Complications in Patients Who Underwent Lung Surgery, Open Thoracic Aortic Repair, Thoracic Endovascular Aortic Repair (TEVAR), and Endovascular Aortic Repair (EVAR). A Retrospective Study
Brief Title: Incidence of Mortality and Complications After Lung Surgery, Open Thoracic Aortic Repair, TEVAR, EVAR.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 798/2564(IRB3)
Record Dates: First submitted 2021-10-02; First posted 2021-10-12 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Morality; Lung Cancer; Aortic Aneurysm; Aortic Dissection
Keywords: Mortality; Major complications; Lung surgery; Open aortic surgery; Thoracic endovascular aortic repair; Endovascular aneurysm repair
MeSH Terms: conditions — Lung Neoplasms; Aortic Aneurysm; Aortic Dissection | interventions — Pulmonary Surgical Procedures; Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Lung surgery: Patients underwent lung surgery.
  Interventions: Procedure: Lung surgery
- Open aortic suregry: Patients underwent open aortic surgery.
  Interventions: Procedure: Open aortic surgery
- Thoracic endovascular aortic repair (TEVAR): Patients underwent TEVAR.
  Interventions: Procedure: TEVAR
- Endovascular aneurysm repair (EVAR): Patients underwent EVAR.
  Interventions: Procedure: EVAR

INTERVENTIONS:
Procedure: Lung surgery — Patients underwent lung surgery including wedge resection, lobectomy, segmentectomy, and pneumonectomy.
  Groups: Lung surgery
Procedure: Open aortic surgery — Patients underwent open thoracic surgery or thoracoabdominal aortic surgery.
  Groups: Open aortic suregry
Procedure: TEVAR — Patients underwent TEVAR.
  Groups: Thoracic endovascular aortic repair (TEVAR)
Procedure: EVAR — Patients underwent EVAR.
  Groups: Endovascular aneurysm repair (EVAR)

SUMMARY:
Lung surgery, open aortic surgery, TEVAR, and EVAR are major operations that carry a higher incidence of perioperative mortality and complications compare to other surgery. The study of the incidence of mortality and complications will help the hospital to benchmark with the others. Also the study of the risk factors of mortality and major complications will help to improve the patients' outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients underwent

* thoracic surgery
* open thoracic aortic surgery
* TEVAR
* EVAR

Exclusion Criteria:

* Emergency lung surgery
* Conversion from TEVAR to open thoracic surgery
* Conversion from EVAR to open aortic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent one of these types of surgery 1) thoracic surgery, 2) open thoracic aortic surgery, 3) TEVAR and 4) EVAR
Sampling Method: Non-Probability Sample
Enrollment: 2224 (Estimated)
Dates: Start 2021-10-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of mortality and major complications after lung surgery | 30 days
  The mortality and major complications (CVS, CNS, RS and others) will be recorded.
Incidence of mortality and major complications after open aortic surgery | 30 days
  The mortality and major complications (CVS, CNS, RS and others) will be recorded.
Incidence of mortality and major complications after TEVAR | 30 days
  The mortality and major complications (CVS, CNS, RS and others) will be recorded.
Incidence of mortality and major complications after EVAR | 30 days
  The mortality and major complications (CVS, CNS, RS and others) will be recorded.

SECONDARY OUTCOMES:
Risk factors of mortality and major complications after lung surgery | 30 days
  To identify risk factors eg. smoking, type of surgery, age, etc.
Risk factors of mortality and major complications after open aortic surgery | 30 days
  To identify risk factors eg. smoking, type of surgery, age, etc.
Risk factors of mortality and major complications after TEVAR | 30 days
  To identify risk factors eg. smoking, diagnosis, age, etc.
Risk factors of mortality and major complications after EVAR | 30 days
  To identify risk factors eg. smoking, age, etc.

OTHER OUTCOMES:
Incidence of postoperative delirium | 30 days
  The patients with postoperative delirium required treatment will be described.
Incidence of low muscle mass | 7 days
  Psoas muscle index will be used for the diagnosis of low muscle mass. Psoas muscle index = both psoas muscle area at L3 (from CT scan) divided by body surface area.
  Cut-off values of sarcopenia
  * Male 68.5 cm2/m2
  * Female 52.5 cm2/m2
Risk factors of postoperative stroke. | 30 days
  To identify risk factors eg. smoking, type of surgery, age, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Mahidol University
Locations (1):
- Anesthesiology Department Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No